CLINICAL TRIAL: NCT04153396
Title: Preemptive Infiltration With Betamethasone and Ropivacaine for Postoperative Pain in Laminoplasty or Laminectomy (PRE-EASE)
Brief Title: Preemptive Infiltration With Betamethasone and Ropivacaine for Postoperative Pain in Laminoplasty or Laminectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY 2019-112-02-1
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Neurosurgery
Keywords: Pain, Postoperative; Betamethasone;; Ropivacaine;; Wound Infiltration; Laminoplasty or Laminectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Treatment Group (Experimental): The local infiltration solution in the treatment group will consist of betamethasone and ropivacaine.
  Interventions: Drug: The Treatment group
- The Control group (Active Comparator): The local infiltration solution in the control group will consist of ropivacaine.
  Interventions: Drug: The Control group

INTERVENTIONS:
Drug: The Treatment group — The local infiltration solution in the treatment group will consist of betamethasone and ropivacaine. For local infiltration, a total of 30 ml solution will be prepared for each group, which will include 0.5ml of compound betamethasone injection(betamethasone propionate 5mg and betamethasone sodium phosphate 2mg per 1ml) added to 14.5ml of saline and 15ml of 1% ropivacaine. The surgeon will perform wound infiltration after induction of anesthesia and before surgery. A total of 10 ml of solution will be injected into each level. The study solution will be injected into the subcutaneous tissue, paravertebral muscles, along with the posterior area around the spinous process, lamina, transverse process and the facet joints, along both sides of the planned incision. The epidural space and intrathecal space will not be infiltrated.
  Arms: The Treatment Group
Drug: The Control group — The local infiltration solution in the control group will consist of ropivacaine. For local infiltration, a total of 30 ml solution will be prepared for each group, which will include 15ml of ropivacaine added to 15 ml of saline for the Control group. The surgeon will perform wound infiltration after induction of anesthesia and before surgery. A total of 10 ml of solution will be injected into each level. The study solution will be injected into the subcutaneous tissue, paravertebral muscles, along with the posterior area around the spinous process, lamina, transverse process and the facet joints, along both sides of the planned incision. The epidural space and intrathecal space will not be infiltrated.
  Arms: The Control group

SUMMARY:
Laminoplasty and laminectomy have been used for decades for the treatment of intraspinal space occupying lesions, spinal stenosis, disc herniation, injuries, etc. After these procedures, patients often experience severe postoperative pain at the surgical site. However, current methods of pain control are mostly insufficient. At present, several pain controlling methods are available, to reduce postoperative pain after laminoplasty or laminectomy. Methods for systemic administration include: oral analgesics, intermittent intravenous, intramuscular injections, patient- controlled intravenous analgesia, etc. However, the aforementioned methods may have a lot of side effects, and are usually used after the occurrence of pain and the analgesic effects are sometimes inadequate. Topical administration options use a lower dose of drugs and therefore have less systemic side effects. Pre-emptive injection of local anesthetics can significantly reduce postoperative pain during rest and movement, however, the analgesic effect is maintained for a relatively short period of time. It is necessary to use more cases to explore the other compatibility of drugs with longer duration of action and stronger analgesic effect. Betamethasone as the stereoisomer of dexamethasone is a long-acting corticosteroid, which has long lasting anti-inflammatory properties. Whether betamethasone combined with local anesthetic for laminoplasty or laminectomy has better short-term and long-term effects than the local anesthetic alone has not been reported yet. Therefore, a prospective, randomized, controlled, blinded-endpoint study is needed to compare the postoperative analgesic efficacy of preemptive wound infilteration of ropivacaine alone and betamethasone plus ropivacaine for laminectomy or laminoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery under general anaesthesia for laminectomy or laminoplasty;
* American Society of Anaesthesiologists (ASA) classification of I or II;
* Age 18 to 64 years;
* Participates with an anticipated full recovery within 2 hours postoperatively.

Exclusion Criteria:

* Patient refusal;
* Participants who cannot use a patient-controlled analgesia (PCA) device and cannot understand the instructions of a Visual Analogue Score (VAS);
* Previous history of spinal surgery;
* Allergy to opioids, betamethasone or ropivacaine;
* Peri-incisional infection;
* History of stroke or a major neurological deficit;
* Trauma, deformity;
* Psychological problems;
* Extreme body mass index (BMI) (< 15 or > 35);
* History of excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks), or use of drugs with confirmed or suspected sedative or analgesic effects;
* Patients using systemic steroids;
* Pregnant or breastfeeding;
* Preoperative Glasgow Coma Scale < 15;
* Participants who have received radiation therapy or chemotherapy preoperatively, or with a high probability to require a postoperative radiation therapy or chemotherapy according to the preoperative imaging.
* Not able to give written informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
The cumulative butorphanol dose during the 48 hours after surgery via the PCA device. | Within 48 hours after the operation
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) device. Participates will be advised to push the analgesic demand button if they feel pain.

SECONDARY OUTCOMES:
The Visual Analogue Scale (VAS) during movement (VASm) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours and 72 hours, and 1 week, 2 weeks, 4 weeks, 6 weeks and 3 months and 6 months after surgery.
  The pain will be assessed by the visual analogue scale (VAS) scores: an 11-point VAS score during movement (VASm) will be recorded (0 indicates no pain, 10 indicates the most severe pain imaginable, a higher score means worse pain)
The Visual Analogue Scale (VAS) at rest (VASr) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours and 72 hours, and 1 week, 2 weeks, 4 weeks, 6 weeks and 3 months and 6 months after surgery.
  The pain will be assessed by the visual analogue scale (VAS) scores: an 11-point VAS score at rest (VASr) will be recorded (0 indicates no pain, 10 indicates the most severe pain imaginable, a higher score means worse pain)
The total times that participants press patient-controlled analgesia button | Within 48 hours after the operation
  The total times that participants press patient-controlled analgesia button including effective presses and ineffective presses.
The first analgesia demand on the PCA device | Within 48 hours postoperatively
  The time from the end of the surgery to the first administration of analgesia via the PCA device
Patient Satisfaction Score (PSS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 4 weeks, 6 weeks, 3 months and 6 months after surgery
  The Patient Satisfaction Score (PSS): 0 for unsatisfactory, and 10 for very satisfied
The Postoperative Nausea and Vomiting (PONV) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  The Postoperative Nausea and Vomiting (PONV) will be measured using an ordinal scale, with 0 indicating no nausea; 1, mild nausea not requiring treatment; 2, nausea requiring treatment; 3, vomiting.
Ramsay Sedation Scale (RSS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  The Ramsay Sedation Scale (RSS): A 6-point scale will be used to assess sedation levels, with 1 indicating agitated, anxious; 2, cooperative; 3, only responds to commands; 4, strong response to glabellar tapping or noisy stimulants; 5, weak response to glabellar tapping or noisy stimulants; 6, no response.
The World Health Organization Quality of Life-BREF (WHOQOL-BREF) scores | At 6 months postoperatively
  The World Health Organization Quality of Life-BREF (WHOQOL-BREF) scores will be used to obtain scores for four domains related to quality of life: physical health (7 items), psychological (6 items), social relationships (3items) and environment (8items). It will also include two stand-alone questions on overall quality of life and satisfaction with health. Each question will be rated on a scale of 1-5 with higher scores signifying better quality of life.
The Oswestry Disability Index (ODI) | Preoperatively and at 4 weeks, 6 weeks and 3 months, 6 months after surgery.
  Functional disability will be assessed by the Oswestry Disability Index. It includes 10 questions about pain and activities of daily living. Each item has five response categories from no pain related disability (0), to the worst possible pain disability (100). The ODI has been reported to be the most widely used and validated outcome measure in spinal surgery.
Patient Scar Assessment and the Observer Scar Assessment Scale (POSAS) | At 6 months postoperatively
  The Patient and Observer Scar Assessment Scale includes subjective symptoms of pain and pruritus and consists of 2 numerical scales: The Patient Scar Assessment Scale and the Observer Scar Assessment Scale. It assesses vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for a scar on a score of 1 (normal skin) to 10 (worst scar imaginable). and it incorporates patient assessments of pain, itching, color, stiffness, thickness, relief and overall opinion. Participants were asked to rate the severity of their scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (very different from normal skin)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Itoh T, Tsuji H. Technical improvements and results of laminoplasty for compressive myelopathy in the cervical spine. Spine (Phila Pa 1976). 1985 Oct;10(8):729-36. doi: 10.1097/00007632-198510000-00007. PMID 3909451
- [Background] Takayasu M, Takagi T, Nishizawa T, Osuka K, Nakajima T, Yoshida J. Bilateral open-door cervical expansive laminoplasty with hydroxyapatite spacers and titanium screws. J Neurosurg. 2002 Jan;96(1 Suppl):22-8. doi: 10.3171/spi.2002.96.1.0022. PMID 11795710
- [Background] Gurbet A, Bekar A, Bilgin H, Ozdemir N, Kuytu T. Preemptive wound infiltration in lumbar laminectomy for postoperative pain: comparison of bupivacaine and levobupivacaine. Turk Neurosurg. 2014;24(1):48-53. doi: 10.5137/1019-5149.JTN.8431-13.0. PMID 24535791
- [Background] Ersayli DT, Gurbet A, Bekar A, Uckunkaya N, Bilgin H. Effects of perioperatively administered bupivacaine and bupivacaine-methylprednisolone on pain after lumbar discectomy. Spine (Phila Pa 1976). 2006 Sep 1;31(19):2221-6. doi: 10.1097/01.brs.0000232801.19965.a0. PMID 16946657
- [Background] Hetland ML, Ostergaard M, Ejbjerg B, Jacobsen S, Stengaard-Pedersen K, Junker P, Lottenburger T, Hansen I, Andersen LS, Tarp U, Svendsen A, Pedersen JK, Skjodt H, Ellingsen T, Lindegaard H, Podenphant J, Horslev-Petersen K; CIMESTRA study group. Short- and long-term efficacy of intra-articular injections with betamethasone as part of a treat-to-target strategy in early rheumatoid arthritis: impact of joint area, repeated injections, MRI findings, anti-CCP, IgM-RF and CRP. Ann Rheum Dis. 2012 Jun;71(6):851-6. doi: 10.1136/annrheumdis-2011-200632. Epub 2012 Feb 1. PMID 22302316
- [Background] Watanabe K, Tokumine J, Yorozu T, Moriyama K, Sakamoto H, Inoue T. Particulate-steroid betamethasone added to ropivacaine in interscalene brachial plexus block for arthroscopic rotator cuff repair improves postoperative analgesia. BMC Anesthesiol. 2016 Oct 4;16(1):84. doi: 10.1186/s12871-016-0251-9. PMID 27716229
- [Background] Cherian MN, Mathews MP, Chandy MJ. Local wound infiltration with bupivacaine in lumbar laminectomy. Surg Neurol. 1997 Feb;47(2):120-2; discussion 122-3. doi: 10.1016/s0090-3019(96)00255-8. PMID 9040811
- [Derived] Shrestha N, Han B, Zhao C, Jia W, Luo F. Pre-emptive infiltration with betamethasone and ropivacaine for postoperative pain in laminoplasty and laminectomy (PRE-EASE): a prospective randomized controlled trial. Int J Surg. 2024 Jan 1;110(1):183-193. doi: 10.1097/JS9.0000000000000821. PMID 37800559
- [Derived] Shrestha N, Wu L, Wang X, Jia W, Luo F. Preemptive Infiltration with Betamethasone and Ropivacaine for Postoperative Pain in Laminoplasty or Laminectomy (PRE-EASE): study protocol for a randomized controlled trial. Trials. 2020 May 5;21(1):381. doi: 10.1186/s13063-020-04308-z. PMID 32370780